CLINICAL TRIAL: NCT03557398
Title: Prospective Clinical Study to Assess the Efficacy and Safety of HYDEAL-D Vaginal Pessaries Application on the Treatment of Vaginal Atrophy in Post-menopause Women
Brief Title: Efficacy and Safety of HYDEAL-D Vaginal Pessaries Application on the Treatment of Vaginal Atrophy in Post-menopause Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QQ53-17-01
Record Dates: First submitted 2018-05-18; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Vulvovaginal Atrophy
Keywords: Hyaluronic acid; Post-menopause

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydeal-D vaginal pessaries (Experimental): Vaginal application of Hydeal-D vaginal pessaries
  Interventions: Device: Hydeal-D vaginal pessaries

INTERVENTIONS:
Device: Hydeal-D vaginal pessaries — One vaginal application of Hydeal-D vaginal pessaries every 3 days to a total of 12 consecutive weeks.
  Other Names: Hyalogyn vaginal pessaries

SUMMARY:
This study evaluates the efficacy and safety of hyaluronic acid derivative based vaginal pessaries for the treatment of symptoms of vulvo-vaginal atrophy in post-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal woman (≥12 months since last spontaneous menstrual period, or having 6 months of spontaneous amenorrhea with serum FSH levels >40 IU/L, or had been surgically postmenopausal for more than 6 months)
* Women between 45 and 75 years of age.
* Vaginal pH ≥5
* Vulvovaginal atrophy with VHI < 15
* At least one of the following symptoms of vulvar and vaginal atrophy, assessed as moderate to severe: vaginal dryness, vaginal and/or vulvar irritation/ itching, dysuria, vaginal pain associated with sexual activity
* Women with active sex lives
* Patients who give written informed consent to participate in the trial

Exclusion Criteria:

* Enrollment in other clinical trials within the previous 1 month.
* Patients in previous treatment with any kind of no-hormonal products for local treatment of vaginal atrophy within 1 week
* Patients in previous treatment with either oral or topical hormonal products within 1 month.
* Patients that present clinical signs of vaginal infections such as trichomonas, candida, and bacterial vaginosis (BV); or history of vulgovaginal contact allergy.
* Patients with acute hepatopathy, embolic disorders, severe primary disease of the kidney and hematopoietic system, and history of malignant tumors.
* Positive history of hypersensitivity hyaluronic acid or to any component of the medical device.
* Women with no active sex lives
* Women who do not give informed consent;
* Any condition in the investigator's opinion not suitable for the inclusion were condition for not eligibility of the patient

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Selection of post-menopausal women with symptoms of vulvovaginal atrophy
Enrollment: 40 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Change of the average score of Vaginal Health Index (VHI) | From baseline to 12 weeks of treatment
  Change of Vaginal Health Index (VHI) calculated on the basis of vaginal elasticity, vaginal fluid volume, vaginal pH, vaginal mucosa epithelial integrity, and vaginal moisture on a scale ranging from 1 (poorest) to 5 (best). VHI assigned score is the sum of subscores and ranges from 5 to 25. A lower score corresponds to a greater atrophy.

SECONDARY OUTCOMES:
Change of the average score of Vaginal Health Index (VHI) | From baseline to 4 weeks of treatment
  Change of Vaginal Health Index (VHI) calculated on the basis of vaginal elasticity, vaginal fluid volume, vaginal pH, vaginal mucosa epithelial integrity, and vaginal moisture on a scale ranging from 1 (poorest) to 5 (best). VHI assigned score is the sum of subscores and ranges from 5 to 25. A lower score corresponds to a greater atrophy.
Change of vaginal pH | From baseline to 4 and 12 weeks of treatment
  The pH values are grouped on a four-point scale and scored respectively: pH lower than 5 = 0; pH between 5 and 5.49 = 1; pH between 5.5 and 6.49 = 2; pH higher than 6.49 =3.
Change of patient's perception of vulvovaginal symptoms | From baseline to 4 and 12 weeks of treatment
  Symptoms associated with vulvovaginal atrophy (dryness, irritation/itching, soreness, dysuria, dyspareunia) are reported on a four-point scale (0=absent, 1=mild, 2=moderate, 3=severe).
Improvement of sexual function through questionnaire Female Sexual Function Index (FSFI) | From baseline to 4 and 12 weeks of treatment
  Female Sexual Function Index (FSFI) questionnaire consists of six domains - desire (two items), arousal (four items), lubrication (four items), orgasm (three items), satisfaction (three items), and pain (three items) - answered on a five-point Likert scale (0, no sexual activity; 1, never/very low; 5, always/very high). A score is calculated for each of the six domains, and the total score is obtained by summing all of the items. Total score ranges from 2 to 36. A lower score corresponds to a greater sexual dysfunction.
Improvement of sexual function through questionnaire Female Sexual Distress Scale-Revised (FSDS-R) | From baseline to 4 and 12 weeks of treatment
  Female Sexual Distress Scale-Revised (FSDS-R) questionnaire consists of 13 items scored on a five-point scale (0, never; 1, rarely; 2, occasionally; 2, frequently; 4, always). The total score is obtained by summing all of the items. Total score ranges from 0 to 52. A higher score corresponds to a greater sexual dysfunction.
Amelioration of the vaginal maturation (VM) index | From baseline to 12 weeks of treatment
  Vaginal maturation (VM) index is calculated quantifying the percentages of parabasal, intermediate, and superficial cells. The following formula is used: VMI = [1(% superficial cells)] + [0.6(% intermediate cells)] + [0.2(% parabasal cells)]. The index ranges from 0% to 100%.The higher the maturation index, the higher the number of mature cells (0%-49%, low stimulation of the vaginal epithelium; 50%-64%, moderate stimulation of the vaginal epithelium; 65%-100%, high stimulation of the vaginal epithelium).
Patient's global assessment of overall satisfaction | 4 and 12 weeks of treatment
  Patient's global assessment (PTGA) is evaluated as the patient's overall satisfaction of the treatment scored on a four grade scale, ranging from 0 to 3 (0= dissatisfied or very dissatisfied, 1= moderately satisfied or satisfied, 2= very satisfied and 3= greatly satisfied). A higher score corresponds to a greater satisfaction.
Local tolerability at the application site | 4 and 12 weeks of treatment
  Local tolerability of the product at the application site is evaluated by both the clinician and the patient independently, through a 5-point scale, ranging from 0 to 5 (1 = excellent (no reaction), 2 = good (small reaction that spontaneously resolves), 3 = moderate (reaction tolerated with difficulty by the subject), 4 = poor (reaction needing interruption of treatment), 5 = bad (serious reaction)). A higher score corresponds to a better tolerability.
Safety of the treatment: Collection of adverse events | 4 and 12 weeks of treatment
  Collection of adverse events emerged as consequence of the product application and any other adverse event occurred during the study

CONTACTS AND LOCATIONS:
Locations (2):
- Slovakia (2):
  - Gynkomed s.r.o., Bratislava
  - ULMUS, s r.o., Hlohovec